CLINICAL TRIAL: NCT04497948
Title: An Open-label, Multiple-dose Study of Acalabrutinib, Co Administered With a Proton-pump Inhibitor, in Participants Hospitalized With COVID-19
Brief Title: Acalabrutinib Study With Best Supportive Care in Participants Hospitalized With COVID-19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Data from the CALAVI Phase II trials for Acalabrutinib in patients hospitalized with COVID-19 did not meet their primary efficacy endpoints.
  Based on this higher management made the decision to prematurely terminate the D822FC00005 PK study.
Sponsor: Acerta Pharma BV (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D822FC00005
Record Dates: First submitted 2020-06-16; First posted 2020-08-04 (Actual); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
Keywords: 2019 novel coronavirus disease; Acalabrutinib; Btk inhibitor
MeSH Terms: conditions — COVID-19 | interventions — acalabrutinib

STUDY DESIGN:
Intervention Model Description: Single group multi dose study. Participants to receive Acalabrutinib + PPI and Best Supportive Care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): Single Arm
  Interventions: Drug: Acalabrutinib

INTERVENTIONS:
Drug: Acalabrutinib — Acalabrutinib (CALQUENCE®) is a covalent BTK inhibitor
  Other Names: CALQUENCE®

SUMMARY:
Study D822FC00005 will investigate the Phamacokinetics, Safety and tolerability of Acalabrutinib suspension when delivered via a nasogastric tube and co-administered with a Proton Pump Inhibitor, in the treatment of COVID-19.

DETAILED DESCRIPTION:
This study is to support the ongoing clinical development of acalabrutinib (CALQUENCE®) in hospitalized COVID-19 patients. Because many COVID-19 patients may be unable to swallow capsules due to respiratory failure (eg, they may require endotracheal intubation for ventilator support and Naso Gastric tube placement), it is important to have a clinically acceptable method to administer acalabrutinib (capsules) via NG tube. Furthermore, many hospitalized patients are placed on high doses of proton pump inhibitors (PPIs) (also commonly known as antacid medication). This study is designed to determine the Pharmaco Kinetics (effect of body/ bodily systems on the drug), safety and tolerability of acalabrutinib suspension, when coadministered with a PPI, in participants with confirmed SARS-CoV-2 infection requiring hospitalization due to respiratory failure, attributable to COVID-19 pneumonia and who have an Nasogastric (NG) tube in place.

ELIGIBILITY:
Inclusion Criteria:

1. Participant or legally authorized representative must be able to understand the purpose and risks of the study and provide written informed consent and authorization to use protected health information (in accordance with national and local patient privacy regulations).
2. Participants who are hospitalized with coronavirus (SARS-CoV-2) infection, confirmed by PCR test or other commercial or public health assay in any specimen, as documented by either of the following:

   1. PCR positive in sample collected < 72 hours prior to first dose, OR
   2. PCR positive in sample collected ≥ 72 hours prior to first dose (but no more than 14 days prior to first dose), documented inability to obtain a repeat sample (eg, due to lack of testing supplies, limited testing capacity, results taking > 24 hours, etc), AND progressive disease suggestive of ongoing SARS-CoV-2 infection 3 Evidence of respiratory failure attributable to COVID-19 pneumonia (documented radiographically) before enrollment 4 Nasogastric tube or other types of oral or percutaneous gastric feeding tube; placement must be radiographically confirmed and expected to remain in place, as judged by the investigator, for a minimum of 3 days after study enrolment.

      5 Has received treatment with PPIs (eg, omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole) for a minimum of 24 hours immediately prior to enrollment; any PPI will be permitted, provided it meets the minimum equivalent daily dose of 20 mg rabeprazole.

      Exclusion Criteria:
      1. Any serious and uncorrectable medical condition or abnormality of clinical laboratory tests that, in the Investigator's judgment, precludes the participant's safe participation in and completion of the study.
      2. In the opinion of the Investigator, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments.
      3. Current refractory nausea and vomiting, malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach, extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
      4. Received BTK inhibitor within 7 days before enrollment.
      5. Requires or is receiving anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon) within 7 days prior to enrollment. Other anticoagulants are permitted.
      6. Participants on dual antiplatelet and therapeutic anticoagulant therapy (eg, aspirin and therapeutic doses of low molecular weight heparin are not allowed; however, aspirin and prophylactic/ low doses of low-molecular-weight heprin are allowed).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D822FC00005&attachmentIdentifier=07a3f757-baee-4846-9350-9804ab60517d&fileName=D822FC005_CSR_Synopsis_redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D822FC00005&attachmentIdentifier=2db78d6d-de17-43c1-bf3e-faab61f41e3a&fileName=D822FC00005_CSP_redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D822FC00005&attachmentIdentifier=e2ace9db-035d-4763-b419-d5522b9ff114&fileName=D822FC00005_SAP_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 20 participants were planned to be enrolled to have at least 16 evaluable participants.
Pre-assignment Details: The study enrollment was terminated early due to the termination of the Calquence COVID-19 Clinical development program (LSPC Nov 2020)
Groups:
- Acalabrutinib + BSC + PPI: Acalabrutinib with Best Supportive Care also with the Proton-Pump Inhibitor(PPI) treatment.
Period: Overall Study
Arm/Group | Acalabrutinib + BSC + PPI
Started | 9
Completed | 7
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Acalabrutinib + BSC + PPI
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (10.7)
Age, Customized [Number; unit: Participants]
  < 65 years | 4
  >= 65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  WHITE | 7
  BLACK OR AFRICAN AMERICAN | 2
  AMERICAN INDIAN OR ALASKA NATIVE | 0
  ASIAN | 0
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 0
  OTHER | 0
  NOT REPORTED | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From 0 to 12 Hours (AUC12h) for Acalabrutinib and ACP-5862 in Visit 1 (Day 1), Visit 2 (Day 2), and Visit 3 (Day 5)
Description: To summarize the PK parameter AUC12h of Acalabrutinib/ACP-5862 in single arm, Acalabrutinib + BSC + PPI
Time Frame: pre-dose and 0.5, 1, 2, 4, 6, and 12 hours in visit 1 on Day 1, visit 2 on Day 2 and visit 3 on Day 5
Population: Here, number analyzed in each row signifies only the participants with available data that were analyzed for each Acalabrutinib and ACP-5862 analytes.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h·ng/mL
Groups:
- Acalabrutinib + BSC + PPI, Visit 1 on Day 1: Acalabrutinib with Best Supportive Care also with the Proton-Pump Inhibitor(PPI) treatment in visit 1 on Day 1.
- Acalabrutinib + BSC + PPI, Visit 2 on Day 2: Acalabrutinib with Best Supportive Care also with the Proton-Pump Inhibitor(PPI) treatment in visit 2 on Day 2.
- Acalabrutinib + BSC + PPI, Visit 3 on Day 5: Acalabrutinib with Best Supportive Care also with the Proton-Pump Inhibitor(PPI) treatment in visit 3 on Day 5.
Arm/Group | Acalabrutinib + BSC + PPI, Visit 1 on Day 1 | Acalabrutinib + BSC + PPI, Visit 2 on Day 2 | Acalabrutinib + BSC + PPI, Visit 3 on Day 5
Number analyzed (Participants) | 9 | 9 | 7
h·ng/mL
  Acalabrutinib | 524.7 (86.5) | 496.5 (58.0) | 201.1 (95.3)
  ACP-5862: number analyzed (Participants) | 8 | 9 | 7
  ACP-5862 | 832.8 (29.3) | 1228.0 (35.1) | 867.1 (43.1)

2. Primary Outcome: Area Under the Concentration-time Curve From 0 to Time to Last Quantifiable Concentration (AUClast) for Acalabrutinib and ACP-5862 in Visit 1 (Day 1), Visit 2 (Day 2), and Visit 3 (Day 5)
Description: To summarize the PK parameter AUClast for Acalabrutinib/ACP-5862 in single arm, Acalabrutinib + BSC +PPI
Time Frame: pre-dose and 0.5, 1, 2, 4, 6, and 12 hours in visit 1 on Day 1, visit 2 on Day 2 and visit 3 on Day5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h·ng/mL
Groups:
- Acalabrutinib + BSC + PPI, Visit 1 on Day 1: Acalabrutinib with Best Supportive Care also with the Proton-Pump Inhibitor(PPI) treatment.
- Acalabrutinib + BSC + PPI, Visit 3 on Day 5: Acalabrutinib with Best Supportive Care also with the Proton-Pump Inhibitor(PPI) treatment on visit 3 on Day 5.
Arm/Group | Acalabrutinib + BSC + PPI, Visit 1 on Day 1 | Acalabrutinib + BSC + PPI, Visit 2 on Day 2 | Acalabrutinib + BSC + PPI, Visit 3 on Day 5
Number analyzed (Participants) | 9 | 9 | 7
h·ng/mL
  Acalabrutinib | 490.1 (64.8) | 493.7 (58.4) | 193.7 (96.6)
  ACP-5862 | 731.0 (38.4) | 1228.0 (35.1) | 827.9 (46.2)

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Acalabrutinib and ACP-5862 in Visit 1 (Day 1), Visit 2(Day2) and Visit 3 (Day 5)
Description: To summarize the PK parameter Cmax of Acalabrutinib/ACP-5862 in single arm, Acalabrutinib + BSC +PPI
Time Frame: pre-dose and 0.5, 1, 2, 4, 6, and 12 hours in visit 1(Day 1), visit 2(Day 2) and visit 3(Day 5)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Acalabrutinib + BSC + PPI, Visit 1 on Day 1 | Acalabrutinib + BSC + PPI, Visit 2 on Day 2 | Acalabrutinib + BSC + PPI, Visit 3 on Day 5
Number analyzed (Participants) | 9 | 9 | 7
ng/mL
  Acalabrutinib | 297.0 (56.7) | 307.9 (51.3) | 167.1 (88.7)
  ACP-5862 | 213.1 (62.9) | 316.9 (38.5) | 324.2 (47.6)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Acalabrutinib + BSC + PPI
All-Cause Mortality (participants affected / at risk) | 2/9
Serious Adverse Events (participants affected / at risk) | 5/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib + BSC + PPI (N=9)
Device related infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 2 (2)
Transaminases increased (Investigations) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib + BSC + PPI (N=9)
Anaemia (Blood and lymphatic system disorders) | 5 (6)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Klebsiella infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Hepatic enzyme increased (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (3)
Polyneuropathy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall provide copies of any materials relating to the Study, or the Developed Technologies that either intends to publish or make any presentations relating to, at least 30 days in advance of publication, submission or presentation.

PI shall not include in or shall remove from any proposed publication of any Confidential Information, errors or inaccuracies; and shall withhold publication, submission for publication or presentation for 90 days from the date the Company receives the material.

DOCUMENTS (2):
  • Study Protocol (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT04497948/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT04497948/SAP_001.pdf